CLINICAL TRIAL: NCT06646484
Title: Interest of Impedancemetry in Monitoring Hydration and Hyponatremia During Subarachnoid Hemorrhages
Acronym: BIASHA
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0783; 2024-A02117-40 (Other: ID-RCB)
Record Dates: First submitted 2024-10-11; First posted 2024-10-17 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Subarachnoid Hemorrhage (SAH)
Keywords: subarachnoid hemorrhage; impedancemetry; hydration
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients hospitalized due to subarachnoid hemorrhages: Each patient eligible for the study hospitalized due to subarachnoid hemorrhages
  Interventions: Diagnostic Test: Impedancemetry evaluation

INTERVENTIONS:
Diagnostic Test: Impedancemetry evaluation — Each patient eligible for the study will, additionally to the standard care, have repeated measure of impedancemetry along their hospital stay ; Theses measure will be compared to the usual measure of hydration and natremia and agreement between clinical status of interest will be discussed.

SUMMARY:
Subarachnoid hemorrhage (SAH) is a rare and serious form of stroke, mainly linked to the rupture of an intracranial aneurysm responsible for bleeding into the meningeal spaces.

The main late serious complication is delayed cerebral ischemia (DCI), resulting in the appearance of new neurological deficits.

Prevention of ICR involves in particular maintaining euvolemia, and early treatment of hyponatremia, itself dependent on the level of volume.

Evaluation of water status and sodium balance is therefore essential. This assessment is complicated and relies on indirect parameters, both clinical and biological.

Impedancemetry, making it possible to measure water volumes and sodium load, could be an aid in the management of blood volume and sodium intake.

ELIGIBILITY:
Inclusion Criteria:

* Adult man, woman
* Hospitalized following Subarachnoid Hemorrhage within 72 hours of bleeding
* Admitted to the neurological intensive care unit for less than 48 hours
* Being able to understand the ins and outs of the study
* Having expressed his non-opposition

Exclusion Criteria:

* Patients under legal protection
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the neurological ICU of Louis Pradel Hospital Lyon in the 72h post subarachnoid hemorrhage.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-21 (Estimated)

PRIMARY OUTCOMES:
Hydration measurements | Every 48 hours during the mean 21 days of stay in the neurological ICU.
  The level of hydration is quantified by the indicator "Hydration of non-fat mass in%" using the impedancemetry. Threshold values for hydration indices are specific to the measurement performed on the patient and depend on their age, gender and body composition data.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon. Neurological ICU, Lyon, France, France

IPD SHARING:
Plan to Share IPD: No